CLINICAL TRIAL: NCT03929484
Title: A Feasibility Study Evaluating a Novel Mask (Nasal Reservoir Cannula) Plus Nasal Cannula vs. Nasal Cannula Alone for Supplemental Oxygen Delivery in the Treatment of Hospitalized Pediatric Patients With Hypoxemia Due to Severe Pneumonia
Brief Title: A Feasibility Study Evaluating a Novel Mask (Nasal Reservoir Cannula)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Per sponsor advice
Sponsor: University of California, San Francisco (Other)
Collaborators: Infectious Diseases Research Collaboration, Uganda (Other); Intellectual Ventures (Unknown); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 16-21217
Record Dates: First submitted 2018-03-02; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Pneumonia Childhood
Keywords: Pneumonia; Hypoxemia; Oxygen therapy; Oxygen mask
MeSH Terms: conditions — Pneumonia; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Each patient will receive oxygen for 1 hour using a novel mask (nasal reservoir cannula) plus standard nasal cannula (Period 1), followed by a 1-hour period of continued use of the standard nasal cannula alone (Period 2).
  Interventions: Device: Nasal reservoir cannula
- Group B (Experimental): Each patient will receive oxygen for 1 hour using a standard nasal cannula alone (Period 1), followed by a 1-hour period of continued use of the novel mask (nasal reservoir cannula) plus standard nasal cannula (Period 2).
  Interventions: Device: Nasal reservoir cannula

INTERVENTIONS:
Device: Nasal reservoir cannula — The experimental oxygen mask (nasal reservoir cannula) fits over a standard nasal cannula. The system is designed to reduce administered oxygen to deliver an equal or higher fraction of inspired oxygen (FiO2) per oxygen delivered (L/min) compared with a standard nasal cannula alone.

SUMMARY:
This study evaluates the addition of a novel mask (nasal reservoir cannula) to a standard nasal cannula during supplemental oxygenation for the treatment of hospitalized pediatric patients with hypoxemia due to severe pneumonia. Half of patients (Group A) will receive oxygen for 1 hour using a novel mask (nasal reservoir cannula) plus standard nasal cannula (Period 1), followed by a 1-hour period of continued use of the standard nasal cannula delivery (Period 2). Half of patients (Group B) will receive oxygen for 1 hour using a standard nasal cannula (Period 1), followed by a 1-hour period of continued use of the novel mask (nasal reservoir cannula) plus standard nasal cannula (Period 2).

DETAILED DESCRIPTION:
Pneumonia is the leading infectious cause of death among children less than 5 years of age. Hypoxemia is a major fatal complication of pneumonia, and the risk of death increases with increasing severity of hypoxemia. Improving oxygen delivery and extending oxygen supplies to children with hypoxemia due to severe pneumonia could reduce mortality in resource-limited settings.

Global Good has developed a low cost oxygen mask (nasal reservoir cannula) to more efficiently deliver oxygen to the pediatric patient by increasing dead space to recapture a portion of expelled oxygen using the spatial distribution of the nasal reservoir cannula volume and length of surface seal. This nasal reservoir cannula fits over a standard nasal cannula (also termed prong). The system is designed to reduce administered oxygen to deliver an equal or higher fraction of inspired oxygen (FiO2) per oxygen delivered (L/min) compared with a standard nasal cannula alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 1 and ≤ 6 years.
2. Severe pneumonia based on WHO criteria
3. SpO2 ≥ 85% and < 94% by pulse oximetry on room air
4. Hospital admission based on clinician judgment
5. Written informed consent from parent(s)/guardian(s) of subjects must be obtained before any study procedure is performed
6. Body weight ≥ 8 kg and ≤ 26 kg

Exclusion Criteria:

1. Hypercapnia (pCO2 > 55 mm Hg or 7.32 kPa) on room air
2. Acidosis / lactic acidosis (pH <7.20 and/or lactate >6 mg/dL) on room air
3. SpO2 < 85% or ≥ 94% by pulse oximetry on room air
4. SICK score > 2.4
5. Hemoglobin < 7 g/dL
6. Facial abnormalities or trauma precluding use of mask and nasal prongs.
7. Requirement of intubation or non-invasive or invasive positive-pressure ventilation
8. Suspected or known pneumothorax
9. Body weight < 8 kg or > 26 kg
10. Hemodynamic instability based on clinician judgment
11. SpO2 < 90% by pulse oximetry on oxygen, measured at the end of the enrollment and before initiation of Period 1

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 1 hour
  Proportion of screened children who were enrolled This will help inform the design of a definitive clinical trial.
Estimated effect of novel mask on amount of oxygen used (compared to standard nasal cannula alone) | 1 hour
  Difference in volume of oxygen used, in liters (from cylinder) Estimation of effect size will help inform the design of a definitive clinical trial.

SECONDARY OUTCOMES:
Protocol adherence | 2 hours
  Proportion of enrolled children who completed the study, per protocol This will help inform the design of a definitive clinical trial.
Oxygen flow | 1 hour
  Average oxygen flow, in liters per minute
Oxygen saturation (SpO2) | 1 hour
  Average continuous oxygen saturation (SpO2) value
PCO2 | End of each period
  PCO2 (capillary blood gas)
pH | End of each period
  pH (capillary blood gas)
Transcutaneous carbon dioxide (tcpCO2) | 1 hour
  Average continuous transcutaneous carbon dioxide (tcpCO2) value

CONTACTS AND LOCATIONS:
Locations (1):
- Mulago Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No